CLINICAL TRIAL: NCT00197548
Title: A Trial of Micronutrients and Adverse Pregnancy Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Wafaie Fawzi, Harvard School of Public of Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD37701
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Pregnancy; Premature Birth; Infant, Low Birth Weight; Pregnancy Outcomes
Keywords: Women; Pregnancy Outcomes; Nutrition; Vitamins; Tanzania; Maternal and Child Health Outcomes
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multivitamins (Active Comparator): Multivitamins-vitamins B-complex, C, and E
  Interventions: Dietary Supplement: Multivitamins-vitamins B-complex, C, and E
- Placebo (Placebo Comparator): Placebo pill
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multivitamins-vitamins B-complex, C, and E — One daily oral dose of 20 mg of B1, 20 mg of B2, 25 mg of B6, 100 mg of niacin, 50 mcg of B12, 500 mg of C, and 30 mg of vitamin E from randomization until delivery. Participants may continue taking this intervention until 18 months post-partum if they are re-randomized to it after delivery.
  Arms: Multivitamins
Dietary Supplement: Placebo — One daily oral dose of a placebo pill taken from randomization until delivery. Participants may continue taking this intervention until 18 months post-partum if they are re-randomized to it after delivery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy of multivitamin supplementation on fetal loss, low birth weight and severe preterm birth in healthy (HIV negative) women.

DETAILED DESCRIPTION:
Fetal loss, low birth weight and preterm birth are major public health problems worldwide, particularly in developing countries. Birth outcomes are also major predictors of child health and survival in infancy and beyond. The purpose of this study is to examine the efficacy of multivitamin supplementation on fetal loss, low birth weight and severe preterm birth in healthy (HIV negative) women. We also aim to determine whether the potentially protective effect of multivitamin supplements on the risks of low birth weight and preterm birth translate into a sustained reduction in infant mortality.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative
* 12-26 weeks gestational age at screening visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8468 (Actual)
Dates: Start 2001-08; Primary Completion 2004-12 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Fetal loss, low birth weight and pre-term birth. | Delivery

SECONDARY OUTCOMES:
Child morbidity and mortality; child growth | 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD,DrPh, Principal Investigator — Harvard School of Public Health (HSPH)

REFERENCES:
- [Result] Fawzi WW, Msamanga GI, Urassa W, Hertzmark E, Petraro P, Willett WC, Spiegelman D. Vitamins and perinatal outcomes among HIV-negative women in Tanzania. N Engl J Med. 2007 Apr 5;356(14):1423-31. doi: 10.1056/NEJMoa064868. PMID 17409323
- [Derived] Wang D, Shahab-Ferdows S, Lweno ON, Hampel D, Method B, Yelverton CA, Nguyen CH, Aboud S, Allen LH, Fawzi WW. The effects of prenatal and postnatal high-dose vitamin B-12 supplementation on human milk vitamin B-12: a randomized, double-blind, placebo-controlled trial in Tanzania. Am J Clin Nutr. 2024 Mar;119(3):730-739. doi: 10.1016/j.ajcnut.2023.07.023. Epub 2023 Nov 30. PMID 38432714
- [Derived] Cliffer I, Darling AM, Madzorera I, Wang D, Perumal N, Wang M, Liu E, Pembe AB, Urassa W, Fawzi WW. Associations of Diet Quality, Socioeconomic Factors, and Nutritional Status with Gestational Weight Gain among Pregnant Women in Dar es Salaam, Tanzania. Curr Dev Nutr. 2023 Feb 4;7(3):100041. doi: 10.1016/j.cdnut.2023.100041. eCollection 2023 Mar. PMID 37181931
- [Derived] Kamenju P, Madzorera I, Hertzmark E, Urassa W, Fawzi WW. Higher Dietary Intake of Animal Protein Foods in Pregnancy Is Associated with Lower Risk of Adverse Birth Outcomes. J Nutr. 2022 Nov;152(11):2546-2554. doi: 10.1093/jn/nxac183. Epub 2022 Aug 18. PMID 36774120
- [Derived] Liu E, Wang D, Darling AM, Perumal N, Wang M, Urassa W, Pembe A, Fawzi WW. Multivitamin Supplementation Is Associated with Greater Adequacy of Gestational Weight Gain among Pregnant Women in Tanzania. J Nutr. 2022 Apr 1;152(4):1091-1098. doi: 10.1093/jn/nxab448. PMID 34964890
- [Derived] Wang D, Natchu UCM, Darling AM, Noor RA, Hertzmark E, Urassa W, Fawzi WW. Effects of prenatal and postnatal maternal multiple micronutrient supplementation on child growth and morbidity in Tanzania: a double-blind, randomized-controlled trial. Int J Epidemiol. 2022 Dec 13;51(6):1761-1774. doi: 10.1093/ije/dyab117. PMID 34151973
- [Derived] Madzorera I, Isanaka S, Wang M, Msamanga GI, Urassa W, Hertzmark E, Duggan C, Fawzi WW. Maternal dietary diversity and dietary quality scores in relation to adverse birth outcomes in Tanzanian women. Am J Clin Nutr. 2020 Sep 1;112(3):695-706. doi: 10.1093/ajcn/nqaa172. PMID 32651998
- [Derived] Quinn MK, Smith ER, Williams PL, Urassa W, Shi J, Msamanga G, Fawzi WW, Sudfeld CR. The Effect of Maternal Multiple Micronutrient Supplementation on Female Early Infant Mortality Is Fully Mediated by Increased Gestation Duration and Intrauterine Growth. J Nutr. 2020 Feb 1;150(2):356-363. doi: 10.1093/jn/nxz246. PMID 31605616
- [Derived] Winje BA, Kvestad I, Krishnamachari S, Manji K, Taneja S, Bellinger DC, Bhandari N, Bisht S, Darling AM, Duggan CP, Fawzi W, Hysing M, Kumar T, Kurpad AV, Sudfeld CR, Svensen E, Thomas S, Strand TA. Does early vitamin B12 supplementation improve neurodevelopment and cognitive function in childhood and into school age: a study protocol for extended follow-ups from randomised controlled trials in India and Tanzania. BMJ Open. 2018 Feb 22;8(2):e018962. doi: 10.1136/bmjopen-2017-018962. PMID 29472265